CLINICAL TRIAL: NCT00904722
Title: Phase II Safety and Efficacy Study of the Monoclonal Antibody CT-011 in Combination With Rituximab in Patients With Relapsed Follicular Lymphoma
Brief Title: Monoclonal Antibody CT-011 in Combination With Rituximab in Patients With Relapsed Follicular Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: CureTech Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009-0163; NCI-2011-03225 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2009-05-18; First posted 2009-05-20 (Estimated); Results first posted 2016-06-03 (Estimated); Last update posted 2016-06-03 (Estimated); Status verified 2016-04

CONDITIONS: Lymphoma
Keywords: Follicular lymphoma; Immunotherapy; CT-011; Monoclonal Antibody CT-011; Rituximab; Rituxan
MeSH Terms: conditions — Lymphoma; Lymphoma, Follicular | interventions — pidilizumab; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CT-011 in combination with Rituximab (Experimental): Combination of the immunotherapy drugs, CT-011 and rituximab.
  Interventions: Drug: CT-011; Drug: Rituximab

INTERVENTIONS:
Drug: CT-011 — Administered intravenously at a dose of 3.0 mg/kg on days 1, 29 (+/- 7 days), 57 (+/- 7 days), and 85 (+/- 7 days).
  Other Names: Monoclonal Antibody CT-011
Drug: Rituximab — Administered intravenously at the standard dose of 375 mg/m^2 weekly for 4 weeks on days 17 (+/- 1 day), 24 (+/- 1 day), 31 (+/- 1 day), and 38 (+/- 1 day).
  Other Names: Rituxan

SUMMARY:
The goal of this clinical research study is to learn if the combination of the immunotherapy drugs, CT-011 and rituximab, can help control follicular lymphoma. The safety of this drug combination will also be studied.

DETAILED DESCRIPTION:
The Study Drugs:

Rituximab is designed to attach to lymphoma cells, which may cause them to die.

CT-011 is designed to strengthen the immune system against cancer, possibly helping the immune cells kill the lymphoma cells better.

Study Drug Administration:

If you are found to be eligible to take part in this study, you will receive an infusion of CT-011 every 4 weeks for a total of 4 infusions. The first infusion will take at least 2 hours and will be given through a needle in your vein. Later infusions will take at least 1 hour. You must stay at the hospital for 2 hours after each infusion. If the lymphoma remains stable or is shrinking after 4 infusions of CT-011, you may receive 8 additional infusions of CT-011 every 4 weeks, for a total of 12 infusions.

You will receive rituximab as an infusion through a needle in your vein once a week for a total of 4 infusions. The first infusion of rituximab will begin about 17 days after the first infusion of CT-011. Each rituximab infusion will be given over 4-8 hours.

You will be watched carefully before, during, and after each CT-011 or rituximab infusion in case you experience any side effects to the drug. You will be given Benadryl (diphenhydramine) and Tylenol (acetaminophen) about 30 to 60 minutes before each infusion in order to lower the risk of possible side effects. If the doctor thinks it is needed, you may also be given other drugs such as hydrocortisone or prednisone (also known as corticosteroids) to help lower the risk of possible side effects. If the side effects become intolerable, and the doctor thinks it is necessary, the infusion may be stopped for a short time or stopped completely.

Study Visits:

The following tests will be performed at your scheduled study visits.

Within 30 days before the first infusion of study drug (up to 2 weeks after the screening tests are complete):

* Blood (about 4 ½ tablespoons) will be drawn for research tests designed to study the function of immune cells in your body.
* Up to 5 needle biopsies (mandatory) will be collected from an enlarged lymph node to collect tumor tissue for research tests. To collect needle biopsies, the area of the tumor is numbed with anesthetic, and a small amount of tumor tissue is withdrawn using a needle.

Blood (about 1 teaspoon each time) will be drawn for research tests to check the levels of CT-011 in the blood and measure how your immune system responds to the drug. These will be drawn right after and then 2 hours after each infusion of CT-011, and on Days 7, 24, 31, 38, and 43.

About 24 hours after the first CT-011 infusion:

-Blood (about 2 ½ tablespoons) will be drawn for research tests to learn if the study drug activates the immune cells.

Before the first rituximab infusion:

* Your medical history will be recorded.
* You will have a physical exam.
* You will have an ECG.
* Blood (about 1 tablespoon) will be drawn for routine tests.
* Blood (about 2 ½ tablespoons) will be drawn for research tests to learn if the study drug activates the immune cells longer than 2 weeks.

Before the second, third, and fourth CT-011 infusion:

* Your medical history will be recorded.
* You will have a physical exam.
* You will have an ECG.
* Blood (about 1 tablespoon) will be drawn for routine tests.
* Blood (about 2 ½ tablespoons) will be drawn for immune-response research tests.

Before the third CT-011 infusion:

* You will have x-rays and CT scans of the neck, chest, abdomen, and pelvis to check the disease status. You may also have a PET scan if your doctor thinks it is needed.
* If your bone marrow was affected by the lymphoma before starting this study, you will have 2 bone marrow biopsies and 1 bone marrow aspirate collected, to check the disease status.

About 4 weeks after the fourth infusion of CT-011:

* Your medical history will be recorded.
* You will have a physical exam.
* You will have an ECG.
* Blood (about 1 tablespoon) will be drawn for routine tests.
* You will have x-rays and CT scans of the neck, chest, abdomen, and pelvis to check the status of your lymphoma. You may also have a PET scan if your doctor thinks it is needed.
* If your bone marrow was affected by lymphoma before starting therapy, you will have 2 bone marrow biopsies and 1 bone marrow aspirate collected to check the status of the disease.
* Blood (about 2 ½ tablespoons) will be drawn for immune-response research studies.

Before CT-011 infusions 5 through 12:

* Your medical history will be recorded.
* You will have a physical exam.
* Blood (about 1 tablespoon) will be drawn for routine tests.

Length of Study:

You may continue receiving CT-011 for up to a total of 12 infusions. You will be taken off study if you have intolerable side effects or the disease gets worse.

Long-Term Follow-Up:

You will be asked to return to the clinic for the following long-term follow-up tests:

About every 3 months after you complete 4 infusions of CT-011:

* Your medical history will be recorded.
* You will have a physical exam.
* You will have an ECG at the final study completion visit.
* Blood (about 1 tablespoon) will be drawn for routine tests.
* You will have x-rays and CT scans of the neck, chest, abdomen, and pelvis to check the disease status.

If your CT scans show that the lymphoma has gone away completely during the above visits, you may also have a PET scan and 2 bone marrow biopsies and 1 bone marrow aspirate collected to confirm the disease status.

At 3, 6, 9, and 12 months after the end of treatment:

-Blood (about 2 ½ tablespoons each time) will be drawn for immune-response research studies.

This is an investigational study. Rituximab is FDA approved and commercially available for the treatment of non-Hodgkin's lymphomas, including follicular lymphoma.

CT-011 is not FDA approved or commercially available. At this time, this drug is being used in research only.

Up to 30 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologic proof of follicular lymphoma grade 1 or grade 2 relapsing after at least 1 but no more than 4 prior systemic therapies.Patients may have had prior local radiation therapy in addition to up to 4 prior systemic therapies. History of total body irradiation will be considered as prior systemic therapy.
2. If patient received prior rituximab-based therapy, should have rituximab sensitive disease defined as a complete or partial response of at least 6 months duration with the rituximab-based regimen.
3. Patients must be >= 18 years of age.
4. Should have measurable (>= 1.5 cm) disease.
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
6. At least 4 weeks from last chemotherapy, immunotherapy, radiation therapy, monoclonal antibody therapy, or experimental therapy and must have recovered from acute toxic effects of prior therapy.
7. Absolute neutrophil count >= 1.5 × 10^9/L.
8. Platelets >= 50 × 10^9/L.
9. Absolute lymphocyte count >= 0.6 × 10^9/L.
10. Adequate renal function with creatinine <= 1.5 × the upper limit of normal (ULN).
11. Adequate hepatic function with total bilirubin <= 1.5 mg/dL; AST and ALT <= 2.5 × ULN.
12. Women of child-bearing potential (i.e., woman has not been naturally postmenopausal for at least 24 consecutive months or not surgically sterile) and sexually active men must agree to use 2 acceptable contraceptive methods during this study. One of the 2 methods of birth control must be a condom. Acceptable methods of birth control in combination with condoms include diaphragm, birth control pills, injections, intrauterine device, and/or under-the-skin implants. Men and women must agree to maintain effective contraception for up to 3 months after the last dose of drug is administered.
13. Patients must sign an informed consent indicating that they are aware of the investigational nature of this study.

Exclusion Criteria:

1. Patients positive for HIV, hepatitis B surface antigen, or hepatitis C antibody.
2. Patients requiring concurrent immunosuppressive therapy are excluded. Inhaled or topical steroids for treating mild to moderate respiratory illnesses, allergies, skin rashes or ocular inflammations are allowed.
3. History of central nervous system (CNS) lymphoma.
4. Active or history of autoimmune disease except Hashimoto's thyroiditis. Patients with type I diabetes mellitus are excluded.
5. Active infection or other serious intercurrent medical illness
6. New York Heart Association Class III or IV disease.
7. Pregnant or nursing.
8. History of allogeneic stem cell transplantation.
9. Other concurrent chemotherapy, radiotherapy, immunotherapy, or investigational therapy
10. Any other malignancy except basal or squamous cell carcinoma of the skin, or cervical carcinoma in situ treated with curative intent. Any cancer from which the patient has been disease free for at least 5 years is permissible.
11. Any underlying medical condition which, in the Principal Investigator's opinion, will make the administration of study drug hazardous or obscure the interpretation of adverse events.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2010-01; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sattva S. Neelapu, MD, Study Chair — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Westin JR, Chu F, Zhang M, Fayad LE, Kwak LW, Fowler N, Romaguera J, Hagemeister F, Fanale M, Samaniego F, Feng L, Baladandayuthapani V, Wang Z, Ma W, Gao Y, Wallace M, Vence LM, Radvanyi L, Muzzafar T, Rotem-Yehudar R, Davis RE, Neelapu SS. Safety and activity of PD1 blockade by pidilizumab in combination with rituximab in patients with relapsed follicular lymphoma: a single group, open-label, phase 2 trial. Lancet Oncol. 2014 Jan;15(1):69-77. doi: 10.1016/S1470-2045(13)70551-5. Epub 2013 Dec 11. PMID 24332512
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: January 08, 2010 to January 05, 2012. All recruitment was done at The University of Texas (UT) MD Anderson Cancer Center.
Pre-assignment Details: Thirty-two patients were enrolled, out of which two patients were ineligible and not treated.
Groups:
- Pidilizumab (CT-011): Combination of the immunotherapy drugs, CT-011 and Rituximab. CT-011: Administered intravenously at a dose of 3.0 mg/kg on days 1, 29 (+/- 7 days), 57 (+/- 7 days), and 85 (+/- 7 days). Rituximab: Administered intravenously at the standard dose of 375 mg/m^2 weekly for 4 weeks on days 17 (+/- 1 day), 24 (+/- 1 day), 31 (+/- 1 day), and 38 (+/- 1 day).
Period: Overall Study
Arm/Group | Pidilizumab (CT-011)
Started | 30
Completed | 29
Not Completed | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | Pidilizumab (CT-011)
Number analyzed (Participants) | 30
Age, Continuous [Median (Full Range); unit: years] | 61 [35 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 17
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: Overall response (OR) rate defined as complete response (CR) + partial response (PR). CR: Complete disappearance of all detectable clinical evidence of disease and symptoms if present before therapy. If a PET scan was positive before therapy, a post-treatment residual mass of any size was deemed a complete response provided that it was PET negative. If response was determined by CT scan criteria, lymph nodes that regressed to less than 1·5 cm were deemed to be complete response. The spleen and/or liver, if considered enlarged before therapy should not be palpable on physical examination and be considered normal size by imaging studies, and nodules related to lymphoma should disappear. PR: At least a 50% decrease in sum of the product of the diameters (SPD) of up to six of the largest dominant nodes or nodal masses. No increase in the size of other nodes, liver, or spleen. Splenic and hepatic nodules must regress by ≥ 50% in their SPD. No new sites of disease should be observed.
Time Frame: Response measured after completion of the second and fourth infusions of CT-011, and every 12 weeks thereafter for 2 years or until relapse.
Population: One patient was withdrawn after one infusion of CT-011 as per the treating physician's decision.
Measure: Number; unit: participants
Arm/Group | Pidilizumab (CT-011)
Number analyzed (Participants) | 29
participants
  Complete Response | 15
  Partial Response | 4

2. Secondary Outcome: Progression-Free Survival
Description: Progression-Free Survival (PFS) was measured from enrollment to disease progression or recurrence or death from any cause.
Time Frame: Measured after completion of the second and fourth infusions of CT-011, and every 12 weeks thereafter for 2 years or until relapse.
Population: One patient was withdrawn after one infusion of CT-011 as per the treating physician's decision.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pidilizumab (CT-011)
Number analyzed (Participants) | 29
months | 18.8 [14.7 to NA] — Distributional assumptions were not available making it not possible to obtain an exact 95% confidence interval for the median.

ADVERSE EVENTS:
Time Frame: Adverse events were captured from Day 1 to 30 days from the last treatment by study drug.
Arm/Group | Pidilizumab (CT-011)
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 30/30
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pidilizumab (CT-011) (N=30)
Anaemia (Blood and lymphatic system disorders) | 14 (14)
Fatigue (General disorders) | 15 (15)
Leucopenia (Blood and lymphatic system disorders) | 11 (11)
Thrombocytopenia (Blood and lymphatic system disorders) | 10 (10)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Neutropenia (Blood and lymphatic system disorders) | 6 (6)
Nausea (Gastrointestinal disorders) | 5 (5)
Sweating (General disorders) | 4 (4)
Neuropathy (Nervous system disorders) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Pain (General disorders) | 5 (5)
Oedema (Blood and lymphatic system disorders) | 4 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 3 (3)
Anorexia (Gastrointestinal disorders) | 3 (3)
Hypotension (Cardiac disorders) | 3 (3)
Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes